CLINICAL TRIAL: NCT06494527
Title: A Randomized, Double-blind, Placebo-controlled, Single/Multiple Ascending Dose, Phase 1 International Multi-center Clinical Study to Evaluate the Safety/Tolerability, Pharmacokinetics/Pharmacodynamics of RG002C0106 Injection in Healthy Adults
Brief Title: A Phase 1 Study to Evaluate the Safety/Tolerability, PK/PD of RG002C0106 Injection in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rigerna Therapeutics Co., Ltd.; Rigerna Therapeutics (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG002C0106-001
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RG002C0106 (Experimental): Randomly enrolled subjects receiving the investigational drug will receive subcutaneous injection for administration
  Interventions: Drug: RG002C0106
- placebo (Placebo Comparator): Randomly enrolled subjects receiving placebo will receive subcutaneous injection for administration
  Interventions: Drug: RG002C0106

INTERVENTIONS:
Drug: RG002C0106 — RG002C0106 is a siRNA drug targeting complement C3 to silence the related gene through the RNA interfering mechanism and inhibit the expression of C3 protein.

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and PK/PD profiles of RG002C0106 injection in healthy adult subjects. The study will be divided into the following parts:

Part A, conducted : SAD stage Part B, conducted: MAD stage

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability and PK/PD profiles of RG002C0106 injection in healthy adult subjects. The study will be divided into the following parts:

Part A, conducted : SAD stage Part B, conducted: MAD stage There are 5 cohorts for the SAD escalation scheme. Dose escalation will start with the planned lowest dose 25mg，and the highest dose will be mainly determined based on the data obtained during the study process.

There are 3 cohorts for the MAD stage .The doses for these 3 cohorts are low dose, medium dose, and high dose, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to communicate well with the investigator, understand and follow trial requirements, voluntarily participate in the trial, understand and sign Informed Consent Form (ICF);
2. Healthy adult subjects aged 18 to 60 years (inclusive), male or female;
3. BMI18-32 kg/m2 ;
4. Subjects who have no current or past medical history of clinically significant diseases of the circulatory system, digestive system, nervous system, respiratory system, and urinary system, mental disorders, or metabolic disorders or history of such disease; and whose physical examination, vital signs, electrocardiogram, chest X-ray or blood test and laboratory tests show normal results or abnormal but not clinically significant results (subject to clinical judgment) at the time of screening.
5. WOCBP must have a negative serum pregnancy test and must not be breastfeeding, lactating or planning pregnancy during the study period.
6. A male subject with a female partner of childbearing potential is eligible to participate if he agrees to use acceptable contraception during the treatment period.
7. Evidence of vaccination (medical record and/or positive antibody test) against Neisseria meningitidis infection (types A, C, W and Y and Group B), Streptococcus pneumoniae, and Haemophilus influenzae type b infection is required before initiation of the investigational drug or placebo.

Exclusion Criteria:

1. Known or persistent mental disorders that require medication intervention and may interfere with the subject's participation in the study.
2. Presence or suspicion of active viral, bacterial, fungal or parasitic infections;
3. History of recurrent or chronic infections;
4. History of epidemic meningococcal infection;
5. History of splenectomy or asplenia;
6. History of complement abnormalities or hereditary complement deficiencies;
7. Any skin conditions and/or tattoos that may interfere with the safety assessment of the injection site, or any relevant history of abdominal scar (surgery, burns, etc.);
8. Subjects who have tested positive for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, and treponema pallidum antibody (optional );
9. Hepatic function abnormal.
10. Renal function abnormal.
11. Allergic condition (allergy to multiple drugs and food) or a known history of allergic reactions to oligonucleotides or hypersensitivity to subcutaneous injections;
12. Subjects who participate in other interventional clinical studies and receive interventional therapy within 30 days before the first dose of the study drug in this study or within the 5 half-lives of the study drug (including investigational drugs and investigational devices) in other interventional clinical studies, whichever is longer.
13. Subjects with history of drug abuse within 12 months.
14. Use of non-prescription drugs within 14 days prior to the first dose of the study drug or within the 5 half-lives of the non-prescription drugs (whichever is longer), unless the investigator determines that the medication is not clinically significant.
15. Subjects who have consumed more than 14 units of alcohol per week.
16. Heavy smoker.
17. Subjects who have donated or lost blood ≥ 480 mL within 3 months.
18. Subjects who have tested positive for pregnancy test; lactating women.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-09 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) related to the investigational drug | up to 169 days
  Incidence of adverse events (AEs) and serious adverse events (SAEs) related to the investigational drug

IPD SHARING:
Plan to Share IPD: No